CLINICAL TRIAL: NCT01401426
Title: Randomized Prospective Trial: Single Port Laparoscopic Vertical Sleeve Gastrectomy Versus Conventional Five Port Laparoscopic Vertical Sleeve Gastrectomy Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCT01401426
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Obesity; Nutrition Disorders; Body Weight
Keywords: overweight; Obesity, Morbid
MeSH Terms: conditions — Obesity; Nutrition Disorders; Body Weight; Overweight; Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Single incision laparoscopic vertical sleeve gastrectomy (Active Comparator): Active Comparator Patients in this group will undergo laparoscopic vertical sleeve gastrectomy through a single periumbilical incision.
  Interventions: Procedure: Laparoscopic vertical sleeve gastrectomy
- Five port laparoscopic vertical sleeve gastrectomy (Active Comparator): Patients in this group will undergo conventional laparoscopic vertical sleeve gastrectomy using 5 small incisions.
  Interventions: Procedure: Laparoscopic vertical sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic vertical sleeve gastrectomy — Laparoscopic vertical sleeve gastrectomy for the treatment of morbid obesity.
  Arms: Single incision laparoscopic vertical sleeve gastrectomy
Procedure: Laparoscopic vertical sleeve gastrectomy — Laparoscopic vertical sleeve gastrectomy
  Arms: Five port laparoscopic vertical sleeve gastrectomy

SUMMARY:
Vertical Sleeve Gastrectomy has been shown to significantly reduce weight and has been approved as a treatment of morbid obesity. The standard laparoscopic operation requires five small incisions for the introduction of instruments and the band into the patient's abdomen. The investigators have developed a technique for performing this operation through a single incision at the belly button. This study compares this method to the conventional 5-incision approach.

ELIGIBILITY:
Inclusion Criteria:

* BMI >40
* ASA I or II

Exclusion Criteria:

* Comorbid cardiac, pulmonary, renal, hepatic disease
* Bleeding disorder
* Previous gastric/esophageal surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 1 month and 1 year

SECONDARY OUTCOMES:
Quality of life | 1 week and 3 months
Peri-Operative Complications | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's Roosevelt Hospital Center, New York, New York, United States